CLINICAL TRIAL: NCT01159405
Title: A Pilot Study of Biodistribution and Dosimetry of 99mTc-Glycopeptide (99mTc-GP) in Patients With Breast Cancer
Brief Title: The Study of Biodistribution and Dosimetry of 99mTc-Glycopeptide(99mTc-GP) in Patients With Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SeeCure LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SeeCure GP-001; NCT01374529 (obsolete NCT alias)
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Glycopeptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 99mTc-GP (Experimental): 99mTc-GP with SPECT/CT imaging & whole body scan.
  Interventions: Radiation: Radiolabeled (99mTc) GP (Glycopeptide)

INTERVENTIONS:
Radiation: Radiolabeled (99mTc) GP (Glycopeptide) — one injection of Technetium Glycopeptide to yield a target activity of 20-25 mCi to be given by slow IV push (over 3-5 minutes) 5 mg, 10 mg & 20 mg of GP will be injected

SUMMARY:
The purpose of this study is to evaluate the biodistribution and dosimetry of single dose of 99mTc-glycopeptide (99mTc-GP, 20-25 mCi) in 3 different doses of GP (5, 10and 20 mg)in patients with breast cancer at pre-chemotherapy.

DETAILED DESCRIPTION:
Cohorts of 3 will be treated each at different dose levels and images will be taken at 4 time points. For dosimetry estimates, there will be a 20-24 hr time point post-administration of 99mTc-GP for the first 3 patients. If the biodistribution and dosimetry can be adequately quantified without the 20-24 hr scan in 3 patients, then we will eliminate that 4th scan for all other patients. Urine and blood samples will be collected at 5 time points, and an additional blood and urine sample will be collected for dosimetry analysis at 30~60 min.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stage I-IV breast cancer (tumor size

  * 2cm in imaging examinations) who are scheduled to start systemic therapy.
* Patients must have histological diagnosis of invasive breast cancer.
* Extent of disease will be determined by physical examination and conventional radiological studies.
* Must be age 18 or older.
* ECOG performance status 0-2.
* Patients with history of prior malignancies must be disease-free for at least 5 years of study entry.
* Normal hematological function: WBC > 3000/ul, absolute neutrophil count > 1500/ul, platelets > 100,000/ul, and Hgb > 10 gms (transfusion to achieve Hgb > 10 gms is acceptable).
* Serum total bilirubin < 1.5 mg/dl and SGPT < 1.5 X normal.
* Adequate kidney function (creatinine < 1.5 mg/dL).

Exclusion Criteria:

* Patients who received previous chemotherapy for the newly diagnosed breast cancer.
* No evidence of primary breast lesion (e.g. T0, Tx).
* Pregnant women or sexually active women of childbearing potential who are not practicing adequate contraception are excluded.
* Patients with myocardial infarction within 6 months of study entry; unstable angina pectoris; uncontrolled congestive heart failure; uncontrolled arrhythmia are excluded.
* Patients with history of hypersensitivity/allergy to Chitosan/Chitin related shellfish foods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
To determine the best dose of 99mTc-GP in imaging based upon safety data and tumor-to background (T/B) count density ratios. | from 99mTc-GP injection through 30 days

SECONDARY OUTCOMES:
To determine the optimal time to imaging after injection of 99mTc-GP based upon tumor to-background (T/B) count density ratios at various times. | from 99mTc-GP injection through 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tejal Patel, M.D., Principal Investigator — Breast Medical Oncologist, Methodist Cancer Center, Houston, Texas
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States